CLINICAL TRIAL: NCT05256589
Title: Clinical Evaluation of the SONA Saliva C-19 Rapid Self-Test for the Detection of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sona Nanotech Inc (Industry)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DHF009 - NSHCT
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Sars-CoV-2 Infection
Keywords: Antigen; COVID19; Rapid Test; Saliva; Self-test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to validate the performance of the Sona Saliva C-19 rapid Self-Test for detection of SARS_CoV_2 infection when using saliva specimens. A prospective study to evaluate a rapid point of care antigen test for the detection of viral proteins and compared against an approved RT-PCR test.
  Saliva samples will be collected along with the current standard of care collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARS_CoV_2 Antigen Rapid Test (Experimental): The same group of patients participate in two arms of the study:
  One arm is for obtaining performance data of the Sona Saliva C-19 Rapid self test and the comparator arm is to obtain data from the primary care route using approved RT-PCR testing.
  Interventions: Diagnostic Test: Sona Saliva C-19 Rapid Self-test

INTERVENTIONS:
Diagnostic Test: Sona Saliva C-19 Rapid Self-test — Rapid Antigen diagnostic device performance comparative to RT-PCR

SUMMARY:
The Sona Saliva C-19 Rapid Self-Test is a lateral flow assay intended for detection of the SARS-CoV-2 virus. Performance of the Sona Saliva C-19 Rapid Test assay will be assessed by comparison to an RT-PCR reference method.

DETAILED DESCRIPTION:
This is a prospective, non-randomized clinical evaluation study being carried out in the intended use population in which fresh saliva samples are collected, tested, and interpreted by lay-users and the results are compared to samples evaluated with an authorized high sensitivity molecular RT-PCR test.

The device to be studied is the Sona Saliva C-19 Rapid Self Test.

Participants will be recruited into the study who present at a NS Health Central Zone COVID-19 PCR testing site for COIVID-19 testing. This study does not involve any additional study visits, and all participants will receive the current standard of care.

Patients will provide their RT-PCR sample as per the established testing processes at the health centre and will receive their results through the standard communication pathway. Self-testing using the Sona assay will be conducted at the COVID -19 testing center by individuals in real time.

The participants will be instructed as to not act on the result of their Sona saliva assay, but rather await the gold standard result of RT-PCR.

A usability questionnaire will also be completed by individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18+ years
2. Presenting at designated NS Health Central Zone COVID-19 PCR testing sites.
3. Receiving a RT-PCR COVID-19 test as per standard of care (nasopharyngeal/mid-turbinate swabs).
4. Unvaccinated, partially vaccinated, fully vaccinated and fully vaccinated-boosted patients
5. Provide written informed consent..
6. Patients may have recently been exposed, in close contact, show no symptoms or may be presenting or have experienced at least one (1) or more signs or symptoms of COVID-19 within ≤ 6 days:

   1. Fever as self-described or measured ≥ 38 °C (100.4°F)
   2. Chills
   3. Cough
   4. Shortness of Breath
   5. Congestion or Runny Nose
   6. Difficulty Breathing
   7. Muscle or Body Aches
   8. Vomiting
   9. Diarrhoea
   10. New loss of sense of taste or smell
   11. General malaise All patients in whom a test result (positive or negative) is obtained from both the RT-PCR testing and Sona Saliva C-19 Rapid Self-test, will be included in the performance analysis.

Exclusion Criteria:

All patients from whom a non-valid result is obtained from either or both the RT-PCR testing and Sona Saliva C-19 Rapid Self-test will be excluded in the analysis for sensitivity and specificity and will be noted as a test error.

Any rapid tests that produced an invalid test result will be noted as a test error and secondary analysis will be conducted on this cohort of patients to understand any underlying causation.

Patients recruited into the study that are recorded to have consumed anything orally within 30 minutes of conducting a rapid self-test, as per the warnings laid out in the IFU, may be excluded from the analysis to mitigate any interference risks relating to test outcome.

Also, the following:

1. Patients unable to provide a saliva sample for rapid testing
2. Patients unable to provide written consent.
3. Patients previously enrolled in the study
4. Patients undergoing treatment currently and/or within the past thirty (30) days of the study with prescription medication to treat novel Coronavirus SARS-CoV-2 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Percent Positive Agreement (Sensitivity) and Negative Percent Agreement (Specificity) | 35 days from last patient enrolment
  Calculate the performance of the Sona Saliva C-19 Rapid Self Test when compared to RT- PCR

CONTACTS AND LOCATIONS:
Locations (1):
- COVID-19 Assessment centre @bayers lake, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No